CLINICAL TRIAL: NCT05724810
Title: Deep rTMS Modulating Insula Synaptic Density and Smoking Behavior in Schizophrenia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stony Brook University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Anissa Abi-Dargham, Distinguished Professor and Chair of Psychiatry, Stony Brook University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1R61DA056423 (NIH)
Record Dates: First submitted 2023-01-27; First posted 2023-02-13 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Schizophrenia; Smoking Cessation; Tobacco Use
Keywords: PET; UCB-J; fMRI; Schizophrenia; Smoking Cessation; Tobacco Use
MeSH Terms: conditions — Schizophrenia; Smoking Cessation; Tobacco Use | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: After enrollment, participants will be randomized between-subjects to active dTMS or sham.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Active and sham cards do not differ in appearance, and both coils are enclosed within the same helmet, enabling double-blind administration.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Active deep transcranial magnetic stimulation (dTMS) (Experimental): Each treatment consists of 60 trains, each lasting 3 sec and interleaved with a 15 sec delay. The entire treatment is delivered over 20 min. The treatment goes for 5 days/week and for a total of 3 weeks.
  Interventions: Device: Active deep transcranial magnetic stimulation (dTMS)
- Sham (Sham Comparator): Active and sham cards do not differ in appearance, and both coils are enclosed within the same helmet, enabling double-blind administration. The same procedure will be done, the only difference is that the sham card does not deliver any stimulation.
  Interventions: Device: Sham dTMS

INTERVENTIONS:
Device: Active deep transcranial magnetic stimulation (dTMS) — First, the investigators will find the position of the right abductor pollicis brevis (APB) motor cortex, finding the minimal motor threshold (MT) required for its activation, which determines the strength of the pulses. After determining the MT, dTMS stimulation is applied 6 cm anterior to the motor "hot spot", at 120% of the MT. The target threshold is built toward gradually. During the first treatment, participants receive stimulation at 100% of the MT. During the second treatment, stimulation intensity increases to 110% of the MT. Beginning at the third treatment and continuing onward, participants receive treatment at 120% of the MT for the course of the treatment.
  Other Names: repetitive transcranial magnetic stimulation (rTMS)
  Arms: Active deep transcranial magnetic stimulation (dTMS)
Device: Sham dTMS — Sham group will go through the same procedure. The only difference is that the sham card does not deliver stimulation.
  Arms: Sham

SUMMARY:
Purpose of the study: Evaluate the effect of deep repetitive transcranial magnetic stimulation (deep rTMS; hereafter abbreviated as "dTMS") on synaptic density measured with positron emission tomography (PET) and the radiotracer [11C]UCB-J. The investigators also seek to link plasticity changes in the regions targeted by the electric field (especially, the insula) to changes in the functioning of insula circuits and behavioral cigarette usage in patients with schizophrenia (SCZ).

Importance of the study: This is the first study designed to directly evaluate the mechanism of action (MOA) of dTMS for smoking disruption in patients with SCZ. Patients with SCZ are a vulnerable population in high, immediate need of new smoking therapeutics for reducing premature morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18-60
2. DSM-5 criteria for schizophreniform, schizophrenia, schizoaffective disorder, or psychotic disorder not otherwise specified (NOS).
3. DSM-5 diagnosis of nicotine use disorder with current daily smoking, and a desire to cut down or quit.
4. Negative urine toxicology (other than cannabis) maintained throughout study participation
5. Fluent English Speaker
6. Capacity for informed consent

Exclusion Criteria:

1. Clinically significant psychopathology other than schizophrenia, schizophreniform, schizoaffective disorder, or psychotic disorder NOS
2. Current or past substance use disorder, except TUD
3. Current use of smoking cessation medications/products
4. Change in schizophrenia medication within 4 weeks
5. Hospitalization in the last 3 months
6. History of suicidal or homicidal tendencies
7. History of epilepsy, stroke, cerebral aneurysm, significant head injury resulting in >10 min loss of consciousness, movement disorder, clinically significant electrolyte abnormalities, or use of clozapine (seizure risks)
8. Pregnancy or lactation (females)
9. Lack of effective birth control (females)
10. Contraindications to MRI or PET
11. Clinical Global Impressions (CGI) rating of 6 (severely ill) or 7 (extremely ill)
12. Prisoners
13. Contraindications to dTMS*

    * The FDA website currently states that the Brainsway device used in this study is contraindicated for patients who have "metallic objects or implanted stimulator devices in or near the head, including cochlear implants, deep brain stimulators, vagus nerve stimulators, other implanted electrodes or stimulators, aneurysm clips or coils, stents, bullet fragments, jewelry and hair barrettes." The investigators will monitor the FDA guidelines and implement any changes to the inclusion/exclusion criteria based on their most updated recommendations.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Estimated)
Dates: Start 2023-04-04 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Insula synaptic density | Change from Baseline at 3 weeks
  PET with UCB-J will be used to look at synaptic density pre/post intervention
Smoking self-administration | Change from Baseline at 3 weeks
  Laboratory tobacco self-administration will be examined pre/post the intervention as a measure of smoking vigor
Insula-centric functional connectivity | Change from Baseline at 3 weeks
  fMRI will be used to look at insula circuit functional connectivity pre/post intervention

SECONDARY OUTCOMES:
Symptoms of Psychosis | up to 4 times over 3 weeks
  The positive and negative syndrome scale (PANSS) will be used to measure symptoms of schizophrenia
Nicotine Craving | post dTMS over 3 weeks
  Craving will be assessed using two self-report items
Cigarettes per Day | Change from Baseline at 3 weeks
  Timeline Follow-back Calendars will be administered pre-dTMS and post-dTMS

CONTACTS AND LOCATIONS:
Locations (1):
- Stony Brook University, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moeller SJ, Gil R, Weinstein JJ, Baumvoll T, Wengler K, Fallon N, Van Snellenberg JX, Abeykoon S, Perlman G, Williams J, Manu L, Slifstein M, Cassidy CM, Martinez DM, Abi-Dargham A. Deep rTMS of the insula and prefrontal cortex in smokers with schizophrenia: Proof-of-concept study. Schizophrenia (Heidelb). 2022 Feb 25;8(1):6. doi: 10.1038/s41537-022-00224-0. PMID 35217662